CLINICAL TRIAL: NCT02789176
Title: Continued Anticonvulsants After Resolution of Neonatal Seizures: a Patient-centered Comparative Effectiveness Study
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: University of California, San Francisco (Other); Boston Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Children's National Research Institute (Other); Massachusetts General Hospital (Other); Patient-Centered Outcomes Research Institute (Other); Stanford University (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Duke University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Renée Shellhaas, MD, Clinical Professor, University of Michigan
Other Study IDs: HUM00114541; 1507-31187 (Other: PCORI project number)
Record Dates: First submitted 2016-05-19; First posted 2016-06-02 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Neonatal Seizures
Keywords: Phenobarbital; EEG; family impact; neurodevelopment
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Outpatient Enrollees: This is a cohort of 150 subjects who were previously enrolled in the Neonatal Seizure Registry, a multi-center association of institutions across the United States, They were contacted to participate in the study after discharge from the Neonatal Intensive Care Unit (NICU) but prior to the prospective follow up. They were asked to take part in all prospective follow up surveys at 12, 18, & 24 months of age.
  Interventions: Other: Surveys
- NICU Enrollees: This is a cohort of 150 subjects who were enrolled in the study prior to discharge from the NICU. They were asked to complete surveys prior to discharge from the NICU, returned to the hospital for a 1 hour EEG to monitor brain activity between 2-4 months of age, & completed the follow surveys at 12, 18, & 24 months of age.
  Interventions: Other: Surveys; Other: EEG

INTERVENTIONS:
Other: Surveys — Regarding development, epilepsy, and family impact
  Other Names: Former Neonatal Seizure Registry Subjects
Other: EEG
  Groups: NICU Enrollees

SUMMARY:
The purpose of this study is to examine whether the duration of treatment with phenobarbital has an impact on neurodevelopmental and epilepsy outcomes, as well as parent and family well-being, after neonatal seizures.

ELIGIBILITY:
Inclusion Criteria:

* Neonates <44 weeks corrected age at seizure onset
* Seizures due to acute brain injury
* Parent(s) who are English or Spanish literate (with assistance of interpreter)

Exclusion Criteria:

* Neonates at risk for adverse outcome independent of seizures and underlying brain injury
* Neonates with mild, temporary causes for seizures
* Newborns with neonatal-onset epilepsy syndromes
* Neonates who do not survive the initial hospital admission
* Neonates will not be excluded based on race, ethnicity, gender or gestational age

Ages: 0 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns with seizures who were admitted at one of the participating children's hospitals
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2016-10; Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renée A Shellhaas, MD, MS, Principal Investigator — University of Michigan; Hannah C Glass, MDCM, MAS, Principal Investigator — University of California, San Francisco
Locations (11):
- United States (11):
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Will be posted on pcori.org

REFERENCES:
- [Derived] Franck LS, Shellhaas RA, Lemmon M, Sturza J, Soul JS, Chang T, Wusthoff CJ, Chu CJ, Massey SL, Abend NS, Thomas C, Rogers EE, McCulloch CE, Grant K, Grossbauer L, Pawlowski K, Glass HC; Neonatal Seizure Registry study group. Associations between Infant and Parent Characteristics and Measures of Family Well-Being in Neonates with Seizures: A Cohort Study. J Pediatr. 2020 Jun;221:64-71.e4. doi: 10.1016/j.jpeds.2020.02.024. PMID 32446494
- See also: PCORI website — http://www.pcori.org/research-results/2016/continued-anticonvulsants-after-resolution-neonatal-seizures-patient-centered

RESULTS

PARTICIPANT FLOW:
Groups:
- Outpatient Enrollees - Maintain Anti-Seizure Medicine: This is a cohort of subjects who were previously enrolled in the Neonatal Seizure Registry and had been discharged from the Neonatal Intensive Care Unit (NICU) on anti-seizure medicine. They were asked to take part in all prospective follow up surveys regarding development, epilepsy, and family impact at 12, 18, & 24 months of age.
- Outpatient Enrollees- Discontinue Anti-Seizure Medicine: This is a cohort of subjects who were previously enrolled in the Neonatal Seizure Registry and had been discharged from the Neonatal Intensive Care Unit (NICU) off anti-seizure medicine. They were asked to take part in all prospective follow up surveys regarding development, epilepsy, and family impact at 12, 18, & 24 months of age.
- Inpatient Enrollees - Maintain Anti-Seizure Medicine: This is a cohort of subjects who were enrolled in the study prior to discharge from the NICU and had been discharged on anti-seizure medicine. They were asked to return to the hospital for a 1 hour EEG to monitor brain activity between 2-4 months of age, and complete surveys regarding development, epilepsy, and family impact prior to discharge from the NICU and at 12, 18, & 24 months of age.
- Inpatient Enrollees - Discontinue Anti-Seizure Medicine: This is a cohort of subjects who were enrolled in the study prior to discharge from the NICU and had been discharged off anti-seizure medicine. They were asked to return to the hospital for a 1 hour EEG to monitor brain activity between 2-4 months of age, and complete surveys regarding development, epilepsy, and family impact prior to discharge from the NICU and at 12, 18, & 24 months of age.
Period: Overall Study
Arm/Group | Outpatient Enrollees - Maintain Anti-Seizure Medicine | Outpatient Enrollees- Discontinue Anti-Seizure Medicine | Inpatient Enrollees - Maintain Anti-Seizure Medicine | Inpatient Enrollees - Discontinue Anti-Seizure Medicine
Started | 99 | 55 | 95 | 54
Completed | 91 | 53 | 85 | 53
Not Completed | 8 | 2 | 10 | 1
Not completed — Death | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 8 | 2 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Outpatient Enrollees - Maintatin Anti-Seizure Medicine: This is a cohort of subjects who were previously enrolled in the Neonatal Seizure Registry and had been discharged from the Neonatal Intensive Care Unit (NICU) on anti-seizure medicine. They were asked to take part in all prospective follow up surveys regarding development, epilepsy, and family impact at 12, 18, & 24 months of age.
- Outpatient Enrollees - Discontinue Anti-Seizure Medicine: This is a cohort of subjects who were previously enrolled in the Neonatal Seizure Registry and had been discharged from the Neonatal Intensive Care Unit (NICU) off anti-seizure medicine. They were asked to take part in all prospective follow up surveys regarding development, epilepsy, and family impact at 12, 18, & 24 months of age.
- Total: Total of all reporting groups
Arm/Group | Outpatient Enrollees - Maintatin Anti-Seizure Medicine | Outpatient Enrollees - Discontinue Anti-Seizure Medicine | Inpatient Enrollees - Maintain Anti-Seizure Medicine | Inpatient Enrollees - Discontinue Anti-Seizure Medicine | Total
Number analyzed (Participants) | 99 | 55 | 95 | 54 | 303
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: Not all subjects completed all the time points and survey questions. Therefore, the number analyzed in the rows may vary.
  Months
    number analyzed (Participants) | 92 | 53 | 79 | 49 | 273
    (all) | 23.89 (0.76) | 23.94 (0.76) | 23.65 (0.56) | 23.97 (0.76) | 23.84 (0.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 26 | 36 | 24 | 133
  Male | 52 | 29 | 59 | 30 | 170
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 6 | 3 | 5 | 6 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 0 | 2
  Black or African American | 12 | 11 | 7 | 6 | 36
  White | 69 | 36 | 59 | 28 | 192
  More than one race | 5 | 0 | 3 | 2 | 10
  Unknown or Not Reported | 7 | 5 | 18 | 11 | 41

OUTCOME MEASURES:

1. Primary Outcome: WIDEA Neurodevelopmental Outcome Score
Description: The Warner Initial Developmental Evaluation of Adaptive and Functional Skills (WIDEA FS) allowed us to compare the functional development between newborns who received short duration phenobarbital treatment and prolonged phenobarbital treatment. There were 50 questions with response options of 1(Never) to 4(all the time). WIDEA range was on a scale from 50-200 (At 24 months, the normal population mean score is 172±10).The higher the score the better the child's developmental function. Mean scores were calculated using data from any participant who completed surveys at 24 months.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Outpatient Enrollees - Maintain Anti-Seizure Medicine | Outpatient Enrollees - Discontinue Anti-Seizure Medicine | Inpatient Enrollees - Maintain Anti-Seizure Medicine | Inpatient Enrollees - Discontinue Anti-Seizure Medicine
Number analyzed (Participants) | 90 | 52 | 79 | 49
score on a scale | 149.04 (34.55) | 162.46 (25.94) | 148.80 (33.52) | 151.89 (33.24)

2. Primary Outcome: Number of Participants With Post-neonatal Epilepsy
Description: The diagnosis of epilepsy and the details of seizure types and frequencies were determined by telephone interview with the parent and corroborated by medical record review.
Time Frame: 24 months
Population: Participants analyzed reflect the number of participants who completed the 24 month follow-up survey. Also one participant did not have data for epilepsy diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Enrollees - Maintain Anti-Seizure Medicine | Outpatient Enrollees - Discontinue Anti-Seizure Medicine | Inpatient Enrollees - Maintain Anti-Seizure Medicine | Inpatient Enrollees - Discontinue Anti-Seizure Medicine
Number analyzed (Participants) | 90 | 53 | 85 | 53
Participants | 14 | 2 | 11 | 10

3. Secondary Outcome: Length of Stay for the Neonatal Seizure Admission
Description: Evaluation of medication exposure (dose and duration) during the admission as a predictor of the number of days the infant requires care (length of stay)
Time Frame: length of stay, measured in days, will be recorded during a chart review when the child is 12 months of age
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Outpatient Enrollees - Maintain Anti-Seizure Medicine | Outpatient Enrollees - Discontinue Anti-Seizure Medicine | Inpatient Enrollees - Maintain Anti-Seizure Medicine | Inpatient Enrollees - Discontinue Anti-Seizure Medicine
Number analyzed (Participants) | 91 | 53 | 85 | 53
number of days | 15 [10 to 25] | 11 [7 to 19] | 17 [9 to 37] | 15 [9 to 31]

4. Secondary Outcome: Impact of Treatment Duration on Parent and Family Well-being
Description: Surveys selected with the help of our Parent Partners were given at 12, 18, and 24 months to assess the impact of neonatal seizure treatment duration on parent and family quality of life and well-being. The 24 month data is presented, as they align with the primary outcome. The study team reviewed the HADS 24 month Anxiety and Depression Score range of possible scores from 0-21 (higher = more depressed/more anxious), the 24 month Transformed WHO Overall Quality of Life and General Health score range of scores 0-100 (higher=better quality of life), the 24 month Impact on Family Scale overall impact scale range from 15-60 (higher = more impact on family), the 24 month Post Traumatic Growth Inventory scale range from 0 -105 (higher = better/more growth), and the 24 month Impact of Events Scale-Revised scale range from 0 - 88 (higher score = worse impact).
Time Frame: 24 months
Population: Not all subjects completed every survey question, therefore some rows have different participants for the various outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Outpatient Enrollees - Maintain Anti-Seizure Medicine | Outpatient Enrollees - Discontinue Anti-Seizure Medicine | Inpatient Enrollees - Maintain Anti-Seizure Medicine | Inpatient Enrollees - Discontinue Anti-Seizure Medicine
Number analyzed (Participants) | 82 | 50 | 70 | 43
score on a scale
  24 month HADS Depression Score | 3.44 (3.01) | 2.92 (2.61) | 3.17 (2.97) | 3.72 (4.04)
  24 month HADS Anxiety Score | 6.15 (4.20) | 5.30 (3.81) | 5.83 (3.79) | 6.84 (4.89)
  24 month Transformed WHO Overall Quality of Life Score: number analyzed (Participants) | 80 | 50 | 60 | 39
  24 month Transformed WHO Overall Quality of Life Score | 76.09 (18.14) | 78.00 (16.67) | 76.67 (17.75) | 75.32 (20.97)
  24 month Impact on Family Scale overall impact scale, 24 mo: number analyzed (Participants) | 81 | 50 | 70 | 43
  24 month Impact on Family Scale overall impact scale, 24 mo | 28.78 (10.41) | 25.50 (9.26) | 28.30 (10.31) | 28.88 (11.42)
  24 month Post Traumatic Growth Inventory | 59.5 (25.1) | 61.9 (25.3) | 61.7 (27.0) | 62.7 (25.0)
  24 month Impact of Events Scale | 15.1 (15.0) | 14.7 (13.6) | 13.8 (13.9) | 16.3 (15.0)

ADVERSE EVENTS:
Time Frame: 24 months
Description: This was an observational study. No intervention was assigned based on participation in the study. All-cause mortality is reported but deaths cannot be attributed to study participation.
Groups:
- Inpatient Enrollees -Discontinue Anti-Seizure Medicine: This is a cohort of subjects who were enrolled in the study prior to discharge from the NICU and had been discharged off anti-seizure medicine. They were asked to return to the hospital for a 1 hour EEG to monitor brain activity between 2-4 months of age, and complete surveys regarding development, epilepsy, and family impact prior to discharge from the NICU and at 12, 18, & 24 months of age.
Arm/Group | Outpatient Enrollees - Maintain Anti-Seizure Medicine | Outpatient Enrollees - Discontinue Anti-Seizure Medicine | Inpatient Enrollees - Maintain Anti-Seizure Medicine | Inpatient Enrollees -Discontinue Anti-Seizure Medicine
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/55 | 3/95 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/55 | 0/95 | 0/54
Other Adverse Events (participants affected / at risk) | 0/99 | 0/55 | 0/95 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT02789176/Prot_SAP_000.pdf